CLINICAL TRIAL: NCT03330977
Title: Efficiency Clinical Study of NOVATEX MEDICAL Compression Garments in Patients With Ehlers-Danlos Syndrome
Acronym: NOVASED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Novatex Medical (Industry)
Collaborators: EVAMED (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-A01531-50
Record Dates: First submitted 2017-10-20; First posted 2017-11-06 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Ehlers-Danlos Syndrome
MeSH Terms: conditions — Ehlers-Danlos Syndrome

STUDY DESIGN:
Intervention Model Description: Comparison before/after
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Before and after use of compression garments (Other): At inclusion, patients will only have medication prescription as usual but without compression garments, and thus, for 4 months.
  4 months after inclusion, patients will continue medication but will also be prescribed compression garments Then every 6 months, until 26 months, patients will come back to have new compression garments (as usual practice)
  Interventions: Device: Compression garments

INTERVENTIONS:
Device: Compression garments — Patients will wear the compression garments since 4 months after inclusion in order to have a comparison before and after use.
  Usual practice would give to the patient the compression garments at inclusion.

SUMMARY:
Objective of this study is to assess the efficiency of NOVATEX MEDICAL compression garments in patients with an Ehlers-Danlos syndrome (EDS).

To answer this objectif a comparison before/after use of compression garments will be performed for all patients.

DETAILED DESCRIPTION:
Inclusion period: 1 year Follow-up period: 26 months Study period : 38 months

Patient visits will be organized as follow:

* V0: first visit at inclusion, clinical evaluation
* V1: 4 months after inclusion, clinical evaluation without compression garments and presure garments prescription
* V2: 8 months after inclusion, clinical evaluation with compression garments
* V3: 14 months after inclusion, clinical evaluation with compression garments
* V4: 20 months after inclusion, clinical evaluation with compression garments
* V5: 26 months after inclusion, clinical evaluation with compression garments

Only the first two visits are specific to the study to be able to compare before and after the use of compression garments. Next visits are the usual visits (every 6 months) for the use of compression garments in patients with an EDS.

ELIGIBILITY:
Inclusion Criteria:

* Patient between 15 and 60 years old
* Ehlers-Danlos Syndrome type: " classical ", " classical-like ", " hypermobile ", " arthrochalasia ", " kyphoscoliotic ", " musculocontractural " ou " myopathic ", as defined in the new international EDS classification 2017
* Patient who have never used compression garments
* Patient for whom compression garments will be prescribed at 4 months
* Patient who have dated and signed a consent form
* Patient who have understood the study
* Patient who are affiliated to French social health insurance system and/or in compliance with the recommendations of the national law in force relating to biomedical research

Exclusion Criteria:

* patient under guardianship or enabled to complete questionnaires
* pregnant or breastfeeding woman
* patient who presents allergy to one of compression garments components
* patient with a current medical history who promotes postural disorders
* patient with an asymptomatic "Hypermobile Sprectrum Disorder" type of EDS as defined in the new international EDS classification 2017
* patient with a current or recent (<3months) participation in another investigational study

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 106 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Improvement of Functional Independence Measure (FIM) scale from 4 months at 8 months | month 4, month 8
  Functional Independence Measure (FIM) is an 18- Item of physical, psychological and social function.
  The FIM uses the level of assistance an individual needs to grade the functional status of a person.
  For each item, disability level is coded from 1 (Total Assistance or not Testable) to 7 (Complete Independence) A total score is calculated using an addition of all items. Thus, score ranges are [18;126]. More the score is high, better is the independence.
  The proportion of patients who present an improvement of 10% of the FIM score between 4 months and 8 months will be calculated.

SECONDARY OUTCOMES:
Patient characteristics | Inclusion
  Describe the characteristics of included patients: age, gender, height, weight, profession, Ehlers-Danlos Syndrom type
Relative improvement of Functional Independence Measure (FIM) scale at 8 months | month 4, month 8
  Functional Independence Measure (FIM) is an 18- Item of physical, psychological and social function.
  The FIM uses the level of assistance an individual needs to grade the functional status of a person.
  For each item, disability level is coded from 1 (Total Assistance or not Testable) to 7 (Complete Independence) A total score is calculated using an addition of all items. Thus, score ranges are [18;126]. More the score is high, better is the independence.
  The FIM score at 8 months will be compared to the FIM score at 4 months.
Evolution of Functional Independence Measure (FIM) scale at long-term from inclusion at 14 months, 20 months and 26 months | Inclusion, month 14, month 20, month 26
  Functional Independence Measure (FIM) is an 18- Item of physical, psychological and social function.
  The FIM uses the level of assistance an individual needs to grade the functional status of a person.
  For each item, disability level is coded from 1 (Total Assistance or not Testable) to 7 (Complete Independence) A total score is calculated using an addition of all items. Thus, score ranges are [18;126]. More the score is high, better is the independence.
  The FIM score will be described at each visit and if relevant, compared to FIM score at inclusion
Evolution of Pain (before and after compression garments using) | Inclusion, month 4, month 8, month 14, month 20, month 26
  Pain evolution using the VAS scale (from 0=no pain to 100=worst imaginable pain) The pain VAS is a continuous scale comprised of a horizontal line, 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme.
  For each visit, proportion of patients who present a decrease of at least 30% of pain score from inclusion, or a pain score <= 2, will be calculated.
Evolution of Tiredness from inclusion at each visit (4 months, 8 months, 14 months, 20 months, 26 months) | Inclusion, month 4, month 8, month 14, month 20, month 26
  Tiredness evolution using Pichot scale Eight items are coded from 0 to 4 (0 = not at all, 1 = a little 2 = moderately 3 = much 4 = extremely).
  Lower is the score, better is the patient tiredness
  For each visit, proportion of patients who present a decrease of at least 30% of Pichot score from inclusion, or a pichot score < 20, will be calculated.
Evolution of Anxiety and depression from inclusion at each visit (4 months, 8 months, 14 months, 20 months, 26 months) | Inclusion, month 4, month 8, month 14, month 20, month 26
  Evolution using the HAD scale (Hospital Anxiety and Depression scale)
  14 items are included in this scale divided in two sub-scores (7 for assessment of the depression and 7 for the assessment of anxiety). A total score is also calculated.
  Lower is the score, better is the patient status
  For each visit, proportion of patients who present a decrease of at least 30% of HAD score from inclusion, or a HAD score < 14, will be calculated.
Evolution of Quality of Life from inclusion at each visit (4 months, 8 months, 14 months, 20 months, 26 months) | Inclusion, month 4, month 8, month 14, month 20, month 26
  Evolution of the Quality of Life using the EQ-5D-3L scale
  This scale is composed of 5 items with 3 levels from 1 to 3.
  Based on these levels, an index can be calculated from 0 to 1. Higher is the score, better is the patient status
  For each visit, proportion of patients who present an improvement of at least 0.10 of index from inclusion will be calculated.
Evolution of the Use of concomitant medication from inclusion at each visit (4 months, 8 months, 14 months, 20 months, 26 months) | Inclusion, month 4, month 8, month 14, month 20, month 26
  Assess the decreasing of use of concomitant medication
  The proportion of patient who present a decreasing of concomitant medication will be calculated at each visit.
Evolution of Compliance | Month 8, month 14, month 20, month 26
  Compliance of compression garments wearing using a patient notebook
  Proportion of patients who are compliant with the compression garments wearing will be calculated at each visit.
  To be compliant is defined by a continuous or daily use
Compression garments safety | month 26
  All adverse events related to the compression garments wearing from inclusion to 26 months will be presented and described
Evolution of Patient satisfaction | month 8, month 14, month 20, month 26
  Patient satisfaction regarding compression garments will be calculated at each visit using the following scale :
  * very satisfied
  * satisfied
  * not satisfied
  * very not satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Roland Jaussaud, Prof., Principal Investigator — Hôpitaux de Brabois - CHRU de Nancy
Locations (10):
- France (10):
  - Centre Médical ISM, Boulogne-Billancourt
  - CHU de CAEN, Caen
  - Hopital Saint Joseph, Marseille
  - Chu de Marseille - Hôpital de La Conception, Marseille
  - Hôpital de L'Hotel Dieu - Aphp, Paris
  - Hopital Lariboisiere, Paris
  - Hopital de La Croix Saint Simon, Paris
  - CHU de REIMS, Reims
  - CHU de SAINT QUENTIN, Saint-Quentin
  - CHRU de NANCY, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No